CLINICAL TRIAL: NCT01184716
Title: The Effect of Vitamin D Fortification of Bread and Milk in Danish Families
Acronym: VitMaD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Denmark (Other)
Responsible Party: Lone Banke Rasmussen, National Food Institute, Technical University of Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 12394
Record Dates: First submitted 2010-08-17; First posted 2010-08-19 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Healthy
Keywords: Vitamin D status (serum 25-hydroxyvitamin D)

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D fortified bread and milk (Active Comparator)
  Interventions: Other: Vitamin D fortification
- Non-fortified bread and milk (No Intervention)

INTERVENTIONS:
Other: Vitamin D fortification — Bread and milk fortified with vitamin D3
  Arms: Vitamin D fortified bread and milk

SUMMARY:
Approximately 200 families corresponding to 800 persons are included in the study. The study investigate the efficacy of vitamin D fortification of bread and milk on vitamin D status in serum. Participants receive milk and bread twice a week. Half of the participants receive vitamin D fortified products and the other half similar non-fortified products. The study starts in September and runs for 6 months during winter, the period where it is not possible to produce vitamin D in the skin through sunlight exposure. The hypothesis is that the usual fall in vitamin D status can be prevented by vitamin D fortified food.

ELIGIBILITY:
Inclusion Criteria:

* Family with at least one child between the age 4 to 18 years and at least one adult less than 60 years of age
* Permanent address in a specific geographical region.

Exclusion Criteria:

* Use of medication (including dietary supplements with high levels of vitamin D)
* Diseases which influence vitamin D metabolism
* Pregnancy

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 782 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxyvitamin D | 6 months
  serum 25-hydroxyvitamin D is measured at the start of the study, after 2-3 months (on adults only) and after approximately 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lone B Rasmussen, M.Sc., Ph.D., Principal Investigator — National Food Institute, DTU
Locations (1):
- Division of Nutrition, National Food Institute, Technical University of Denmark, Søborg, Denmark

REFERENCES:
- [Derived] Nissen J, Vogel U, Ravn-Haren G, Andersen EW, Madsen KH, Nexo BA, Andersen R, Mejborn H, Bjerrum PJ, Rasmussen LB, Wulf HC. Common variants in CYP2R1 and GC genes are both determinants of serum 25-hydroxyvitamin D concentrations after UVB irradiation and after consumption of vitamin D(3)-fortified bread and milk during winter in Denmark. Am J Clin Nutr. 2015 Jan;101(1):218-27. doi: 10.3945/ajcn.114.092148. Epub 2014 Nov 5. PMID 25527766